CLINICAL TRIAL: NCT01559272
Title: A Single-Dose, Open-Label, Randomized, Parallel-Group Study to Assess the Pharmacokinetics, Safety, and Tolerability of a Paliperidone Palmitate 3-Month Formulation in Subjects With Schizophrenia
Brief Title: A Study to Assess the Pharmacokinetics, Safety, and Tolerability of Paliperidone Palmitate in Patients With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR012652; R092670PSY1005 (Other: Janssen Research & Development, LLC); 2007-003581-17 (EudraCT Number)
Record Dates: First submitted 2012-03-13; First posted 2012-03-21 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone palmitate; R092670; Paliperidone; 3-month formulation; Pharmacokinetics
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (4):
- Panel A (Experimental): Panel A consists of 2 treatment groups
  Interventions: Drug: Paliperidone IR (Period 1); Drug: Paliperidone palmitate F015 (Panel A: treatment group 1); Drug: Paliperidone palmitate F015 (Panel A: treatment group 2)
- Panel B (Experimental): Panel B consists of 5 treatment groups
  Interventions: Drug: Paliperidone IR (Period 1); Drug: Paliperidone palmitate F015 (Panel B: treatment group 1); Drug: Paliperidone palmitate F015 (Panel B: treatment group 2); Drug: Paliperidone palmitate F015 (Panel B: treatment group 3); Drug: Paliperidone palmitate F015 (Panel B: treatment group 4); Drug: Paliperidone palmitate F015 (Panel B: treatment group 5)
- Panel C (Experimental): Panel C consists of 1 treatment group
  Interventions: Drug: Paliperidone IR (Period 1); Drug: Paliperidone palmitate F016
- Panel D (Experimental): Panel D consists of 4 treatment groups
  Interventions: Drug: Paliperidone IR (Period 1); Drug: Paliperidone palmitate F015 (Panel D: treatment group 1); Drug: Paliperidone palmitate F015 (Panel D: treatment group 2); Drug: Paliperidone palmitate F015 (Panel D: treatment group 3); Drug: Paliperidone palmitate F015 (Panel D: treatment group 4)

INTERVENTIONS:
Drug: Paliperidone IR (Period 1) — Type= exact number, unit= mg, number=1, form= injection, route= intramuscular use. Single injection with 1 mg paliperidone IR in the gluteal or deltoid muscle.
Drug: Paliperidone palmitate F015 (Panel A: treatment group 1) — Type= exact number, unit= mg, number=300, form= injection, route= intramuscular use. Single injection with 300 mg eq. 3-month formulation paliperidone palmitate F015 manufactured by milling technique A, in the gluteal muscle.
  Arms: Panel A
Drug: Paliperidone palmitate F015 (Panel A: treatment group 2) — Type= exact number, unit= mg, number=300, form= injection, route= intramuscular use. Single injection with 300 mg eq. 3-month formulation paliperidone palmitate F015 manufactured by milling technique B, in the gluteal muscle.
  Arms: Panel A
Drug: Paliperidone palmitate F015 (Panel B: treatment group 1) — Type= exact number, unit= mg, number= 75, form= injection, route= intramuscular use. Single injection with 75 mg eq. 3-month formulation paliperidone palmitate F015 in the gluteal muscle.
  Arms: Panel B
Drug: Paliperidone palmitate F015 (Panel B: treatment group 2) — Type= exact number, unit= mg, number=150, form= injection, route= intramuscular use. Single injection with 150 mg eq. 3-month formulation paliperidone palmitate F015 in the gluteal muscle.
  Arms: Panel B
Drug: Paliperidone palmitate F015 (Panel B: treatment group 3) — Type= exact number, unit= mg, number=450, form= injection, route= intramuscular use. Single injection with 450 mg eq. 3-month formulation paliperidone palmitate F015 in the gluteal muscle.
  Arms: Panel B
Drug: Paliperidone palmitate F015 (Panel B: treatment group 4) — Type= exact number, unit= mg, number=300, form= injection, route= intramuscular use. Single injection with 300 mg eq. 3-month formulation paliperidone palmitate F015 in the deltoid muscle.
  Arms: Panel B
Drug: Paliperidone palmitate F015 (Panel B: treatment group 5) — Type= exact number, unit= mg, number=450, form= injection, route= intramuscular use. Single injection with 450 mg eq. 3-month formulation paliperidone palmitate F015 in the deltoid muscle.
  Arms: Panel B
Drug: Paliperidone palmitate F016 — Type= exact number, unit= mg, number=150, form= injection, route= intramuscular use. Single injection with 150 mg eq. 3-month formulation paliperidone palmitate F016 in the gluteal muscle.
  Arms: Panel C
Drug: Paliperidone palmitate F015 (Panel D: treatment group 1) — Type= exact number, unit= mg, number=525, form= injection, route= intramuscular use. Single injection with 525 mg eq. 3-month formulation paliperidone palmitate F015 in the gluteal muscle.
  Arms: Panel D
Drug: Paliperidone palmitate F015 (Panel D: treatment group 2) — Type= exact number, unit= mg, number=525, form= injection, route= intramuscular use. Single injection with 525 mg eq. 3-month formulation paliperidone palmitate F015 in the deltoid muscle.
  Arms: Panel D
Drug: Paliperidone palmitate F015 (Panel D: treatment group 3) — Type= exact number, unit= mg, number=350, form= injection, route= intramuscular use. Single injection with 350 mg eq. 3-month formulation paliperidone palmitate F015 in the gluteal muscle.
  Arms: Panel D
Drug: Paliperidone palmitate F015 (Panel D: treatment group 4) — Type= exact number, unit= mg, number=175, form= injection, route= intramuscular use. Single injection with 175 mg eq. 3-month formulation paliperidone palmitate F015 in the deltoid muscle.
  Arms: Panel D

SUMMARY:
The purpose of this study is to assess the pharmacokinetics, safety, and tolerability of a paliperidone palmitate 3-month formulation in patients with schizophrenia.

DETAILED DESCRIPTION:
This is a multicenter, randomized (the study drug is assigned by chance), open-label (all people know the identity of the intervention), parallel-group (each group of patients will be initiated simultaneously) study in 4 panels (A, B, C and D). Each panel will comprise 2 single-dose treatment periods. In Period 1, all patients from the 4 panels will receive an intramuscular (i.m.) injection with 1 mg paliperidone as an immediate release (IR) solution to assess tolerability and allergic or hypersensitivity reactions potentially related to paliperidone, and to establish the relative bioavailability (the extent to which a drug or other substance becomes available to the body) of paliperidone palmitate versus paliperidone IR. Patients in Panels A and C will receive an i.m. injection with 1 mg paliperidone IR solution in the gluteal muscle, and patients in Panel B and D will receive an i.m. injection with 1 mg paliperidone IR solution in the deltoid or gluteal muscle. Patients who tolerate this injection and have completed all assessments on Day 5 of Period 1 will be enrolled in Period 2. In Period 2, patients will receive a single dose of 3-month paliperidone palmitate i.m. injection at the dosages defined for each panel. The study drug injection will be followed by a 96-hour observation period in Period 1, and a 364-day or 544-day observation period in Period 2. Successive study drug administrations will be separated by a washout period (period when receiving no treatment) of at least 7 and no more than 21 days. The total study length for all patients is from 53 weeks to a maximum of 58 weeks. Patients in Panel B, if consented, and Panel D will participate in the extension period of approximately 26 weeks in order to obtain additional assessments to be able to characterize the pharmacokinetics (PK) profile. Pharmacokinetics explores how the drug is absorbed in the body, distributed within the body, and how it is removed from the body over time. Therefore, for those who participate in the extension period, the total study duration will be approximately 84 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with schizophrenia or schizoaffective disorder, for at least 1 year before screening
* Clinically stable with no hospitalizations for schizophrenia exacerbation or change in current antipsychotic medications for 3 months prior to screening
* Stabilized on antipsychotic medications other than risperidone, paliperidone, ziprasidone, clozapine, thioridazine, or any long acting injectable.
* For panel D only, no detectable plasma concentration of risperidone or paliperidone > 0.1ng/mL at screening. A quantifiable and stable level of paliperidone not exceeding 0.25 ng/mL is allowed if such paliperidone value is explained by (documented) use of paliperidone palmitate (last dose administered > 12 months prior to baseline)
* Has a total PANSS score of 70 or less at both screening and Day-1 (Period 1)
* Woman is postmenopausal, surgically sterile, abstinent or, if sexually active, practices an effective method of birth control during participation in the study or for at least 6 months after the last dose of study drug, whichever is longer
* Woman has negative pregnancy test at screening and on Day -1 of Period 1
* Man agrees to use an adequate contraception method as deemed appropriate by the investigator and agrees to not donate sperm during participation in the study or for at least 6 months after the last dose of study drug, whichever is longer
* Body Mass Index (BMI) between 17 and 35 kg/m2 (inclusive). Body weight of at least 50 kg for patients enrolled in panel A, B and C. For patients enrolled in panel D only: body weight of at least 47 kg

Exclusion Criteria:

* Attempted suicide within 12 months before screening or is at imminent risk of suicide or violent behavior
* Has diagnosis of alcohol or substance dependence, with the exception of nicotine or caffeine dependence, within 12 months prior to screening, or diagnosis of substance abuse within 3 months prior to screening
* Has a positive drug screen test for barbiturates, cocaine, amphetamines or opiates, or has a positive alcohol screen test unless positive toxicology screen is explained by a prescribed allowed medication
* Is in his/her first episode of psychosis
* Has a history of or has a current clinically significant medical illness that the investigator considers should exclude the patients or that could interfere with the interpretation of the study results
* Has clinically significant abnormal values at screening or at baseline for hematology, clinical chemistry or for urinalysis, as deemed appropriate by the investigator
* Has a clinically relevant abnormality in the physical examination, vital signs or 12 lead electrocardiogram (ECG) at screening or at baseline as deemed appropriate by the investigator
* Has a history or presence of circumstances that may increase the risk of the occurrence of torsade de pointes and/or sudden death in association with the use of drugs that prolong the QTc interval
* Concomitant use of medications that the investigator considers should exclude the patients or that could interfere with the interpretation of the study results
* Any other condition or circumstance that the investigator considers should exclude the patients or that could interfere with the interpretation of the study results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2008-02-21 (Actual); Primary Completion 2014-04-09 (Actual); Study Completion 2014-05-24 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of Paliperidone (Period 1) | 14 time points over 96 hours
Plasma concentration of Paliperidone (Period 2) | 29 time points over 544 days

SECONDARY OUTCOMES:
The change from baseline in Positive and Negative Syndrome Scale for Schizophrenia (PANSS) (Period 1) | Baseline and 96 hours
  The PANSS is a 30-item scale (range 30-210) designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items. Higher scores indicate worsening.
Changes in Positive and Negative Syndrome Scale for Schizophrenia (PANSS) observed across multiple time points between baseline and 544 days (Period 2) | Baseline and 544 days
  The PANSS is a 30-item scale (range 30-210) designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items. Higher scores indicate worsening.
The change from baseline in Clinical Global Impression (CGI-S) (Period 1) | Baseline and 96 hours
  The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a subject. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill subjects". Higher scores indicate worsening.
Changes in Clinical Global Impression (CGI-S) observed across multiple time points between baseline and 544 days (Period 2) | Baseline and 544 days
  The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a subject. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill subjects". Higher scores indicate worsening.
Changes from Baseline in Abnormal Involuntary Movement Scale (AIMS) for the ratings of dyskinesia (Period 1) | Baseline and 96 hours
  The AIMS consists of 12 items to measure involuntary movements known as dyskinesia, with scores ranging from 0 (none) to 4 (severe).
Changes in Abnormal Involuntary Movement Scale (AIMS) for the ratings of dyskinesia observed across multiple time points between baseline and 544 days (Period 2) | Baseline and 544 days
  The AIMS consists of 12 items to measure involuntary movements known as dyskinesia, with scores ranging from 0 (none) to 4 (severe).
Changes from Baseline in Barnes Akathisia Rating Scale (BARS) for the ratings of akathisia (Period 1) | Baseline and 96 hours
  The BARS is a scale to assess the presence and severity of drug-induced akathisia (inner restlessness). It is scored as follows: Objective Akathisia, Subjective Awareness of Restlessness and Subjective Distress Related to Restlessness are rated on a 4-point scale from 0 (normal or absence of restlessness) to 3 (intense restlessness). The Global Clinical Assessment of Akathisia uses a 6-point scale ranging from 0 (absent) to 5 (severe akathisia).
Changes in Barnes Akathisia Rating Scale (BARS) for the ratings of akathisia observed across multiple time points between baseline and 544 days (Period 2) | Baseline and 544 days
  The BARS is a scale to assess the presence and severity of drug-induced akathisia (inner restlessness). It is scored as follows: Objective Akathisia, Subjective Awareness of Restlessness and Subjective Distress Related to Restlessness are rated on a 4-point scale from 0 (normal or absence of restlessness) to 3 (intense restlessness). The Global Clinical Assessment of Akathisia uses a 6-point scale ranging from 0 (absent) to 5 (severe akathisia).
Changes from Baseline in Simpson and Angus Rating Scale (SAS) for the ratings of general extrapyramidal symptoms (EPS) (Period 1) | Baseline and 96 hours
  The SAS is a 10-item instrument used to evaluate the presence and severity of extrapyramidal symptoms (EPS), such as akinesia (inability to initiate movement) and akathisia. Items are rated for severity on a 0 (normal) to 4 (severe symptoms) scale.
Changes in Simpson and Angus Rating Scale (SAS) for the ratings of general extrapyramidal symptoms (EPS) observed across multiple time points between baseline and 544 days (Period 2) | Baseline and 544 days
  The SAS is a 10-item instrument used to evaluate the presence and severity of extrapyramidal symptoms (EPS), such as akinesia (inability to initiate movement) and akathisia. Items are rated for severity on a 0 (normal) to 4 (severe symptoms) scale.
Changes from Baseline in Columbia-Suicide Severity Rating Scale (C-SSRS) (Period 1) | Baseline and 96 hours
  The Columbia-Suicide Severity Rating Scale (C-SSRS) rates an individual's degree of suicidal ideation on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent."
Changes in Columbia-Suicide Severity Rating Scale (C-SSRS) observed across multiple time points between baseline and 544 days (Period 2) | Baseline and 544 days
  The Columbia-Suicide Severity Rating Scale (C-SSRS) rates an individual's degree of suicidal ideation on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent."
Evaluation of the Injection Site (Period 1) | 96 hours
  The investigator will evaluate the site of injection for redness, swelling, and induration. The evaluation will be assessed as 0 = absent, 1 = mild, 2 = moderate, 3 = severe.
Evaluation of the Injection Site (Period 2) | Baseline through day 112
  The investigator will evaluate the site of injection for redness, swelling, and induration. The evaluation will be assessed as 0 = absent, 1 = mild, 2 = moderate, 3 = severe.
Incidence of Adverse Events as a Measure of Safety and Tolerability | Approximately 84 weeks
Number of patients with abnormal clinical laboratory tests | Approximately 84 weeks
Number of patients with abnormal findings in electrocardiogram, vital signs and physical examination | Approximately 84 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (36):
- United States (10):
  - Little Rock, Arkansas
  - Cerritos, California
  - Garden Grove, California
  - Glendale, California
  - National City, California
  - Paramount, California
  - Atlanta, Georgia
  - Philadelphia, Pennsylvania
  - Austin, Texas
  - DeSoto, Texas
- Belgium (2):
  - Aalst
  - Diest
- Burgas, Bulgaria
- Zagreb, Croatia
- Israel (3):
  - Beer Yaakov
  - Hod HaSharon
  - Ramat Gan
- Malaysia (3):
  - Johor Bahru
  - Kuala Lumpur
  - Perak
- Slovakia (3):
  - Bratislava
  - Michalovce
  - Rimavská Sobota
- South Africa (2):
  - Bloemfontein
  - Cape Town
- South Korea (3):
  - Incheon
  - Jeonju
  - Seoul
- Spain (5):
  - Badajoz
  - Badalona
  - Barcelona
  - Seville
  - Zamora
- Taiwan (3):
  - Hualien City
  - Taipei
  - Taoyuan District

REFERENCES:
- [Derived] Magnusson MO, Samtani MN, Plan EL, Jonsson EN, Rossenu S, Vermeulen A, Russu A. Population Pharmacokinetics of a Novel Once-Every 3 Months Intramuscular Formulation of Paliperidone Palmitate in Patients with Schizophrenia. Clin Pharmacokinet. 2017 Apr;56(4):421-433. doi: 10.1007/s40262-016-0459-3. PMID 27743205
- [Derived] Samtani MN, Nandy P, Ravenstijn P, Remmerie B, Vermeulen A, Russu A, D'hoore P, Baum EZ, Savitz A, Gopal S, Hough D. Prospective dose selection and acceleration of paliperidone palmitate 3-month formulation development using a pharmacometric bridging strategy. Br J Clin Pharmacol. 2016 Nov;82(5):1364-1370. doi: 10.1111/bcp.13050. Epub 2016 Jul 24. PMID 27333588
- [Derived] Gopal S, Vermeulen A, Nandy P, Ravenstijn P, Nuamah I, Buron Vidal JA, Berwaerts J, Savitz A, Hough D, Samtani MN. Practical guidance for dosing and switching from paliperidone palmitate 1 monthly to 3 monthly formulation in schizophrenia. Curr Med Res Opin. 2015 Nov;31(11):2043-54. doi: 10.1185/03007995.2015.1085849. Epub 2015 Oct 2. PMID 26306819
- See also: A Single-Dose, Open-Label, Randomized, Parallel-Group Study to Assess the Pharmacokinetics, Safety, and Tolerability of a Paliperidone Palmitate 3-Month Formulation in Subjects With Schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=1916&filename=CR012652_CSR.pdf